CLINICAL TRIAL: NCT06951178
Title: Unlocking TMJs Clinical Study: Safety and Performance of Materialise's Patient-specific TMJ System
Brief Title: Long-term Safety and Performance of Materialise's Patient-specific TMJ System.
Status: Not yet recruiting | Type: Observational
Sponsor: Materialise (Industry)
Responsible Party: Sponsor
Other Study IDs: SMAT013
Record Dates: First submitted 2025-04-14; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Joint Disorders; Implant
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TMJ Total Arthroplasty System (TMJ System) — All patients treated or to be treated with the TMJ Total Arthroplasty System for TMJ reconstruction. The TMJ Total Arthroplasty System (TMJ System) is a medical device intended to restore the TMJ. It comprises two articulating components: a temporal component and a mandibular component. The TMJ System is patient-specific based on the patient's anatomy and surgical treatment. Different shape designs are possible depending on the patient's anatomy and the type of surgery performed.
  Other Names: Temporomandibular joint reconstruction

SUMMARY:
This is a long-term (10 years), retrospective-prospective, observational, single-arm, monocenter study of patients to be treated with the Materialise TMJ Total Arthroplasty System for TMJ replacement. The study will evaluate the efficiency, safety, clinical performance, accuracy, benefits, and risks associated with long-term use and the impact on life quality and diet of the TMJ system, its fixation devices, TMJ Implant trial, and guides in the adolescent and adult populations.

DETAILED DESCRIPTION:
The study begins with patient inclusion and pre-operative examination, where eligibility is assessed based on inclusion and exclusion criteria. Informed consent is obtained, and if a participant drops out before implantation, a new patient is enrolled. Pre-operative assessments include (CB)CT imaging, collection of demographic details, medical history, and co-morbidities using the Charlson Comorbidity Index (CCI). Other pre-operative evaluations include maximal inter-incisal opening (MIO), occlusion, diet consistency, and several questionnaires to assess quality of life, jaw function, and speech. Pre-operative (CB)CT scans are used for surgical planning and device design.

During surgery and hospital stay, the index procedure marks the patient's enrollment. Surgical details are documented, including the approach, device characteristics, operation time, and complications. Intraoperative adverse events, such as allergic reactions or hematoma, are recorded. A post-operative (CB)CT scan is performed within a week, and patient and surgeon satisfaction, both functional and aesthetic, are recorded. Any post-operative complications are tracked.

For follow-up, the study includes 9 follow-up visits at intervals of 1 week, 4 weeks, 3 months, 6 months, 1 year, 2 years, 3 years, 5 years, and 10 years. At each visit, MIO, occlusion, diet consistency, and jaw function are assessed, and patients complete the EQ-5D-5L, OHIP-14, and Helkimo Clinical Dysfunction Index questionnaires. A (CB)CT scan is performed at specific follow-ups, and any post-operative complications, adverse events, or re-interventions are reported. Medication intake is recorded as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed with Materialise TMJ Total Arthroplasty System for TMJ reconstruction
* Patient who has received and understood the study information leaflet and has agreed to participate in the study and signed the informed consent form (ICF) (adult or legal guardian(s) if minor).

Exclusion Criteria:

* Known hypersensitivity to Titanium, Nickel, or Cobalt-Chrome alloys.
* Patient conditions where there is not enough bone quality or quantity to support the components.
* Active infection in the anatomical area or the vicinity of the site to be implanted, preventing the implantation of the device.
* Patients with marked hyperfunctional habits (e.g., tooth clenching, bruxism).
* Pregnant woman.
* Patient is known to be or suspected of being unable to comply with the study protocol or proposed follow-up visits by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated or to be treated with the Materialise TMJ Total Arthroplasty System for TMJ reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2037-06 (Estimated); Study Completion 2037-06 (Estimated)

PRIMARY OUTCOMES:
Implant success rate | 10-year follow-up post-implantation, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  This metric evaluates the percentage of implanted devices that remain in place and functional over a 10-year follow-up period. It directly reflects the device's safety and long-term effectiveness. Success in durability is defined as device securely in place and functional at 10-year follow-up given implant stability & joint function. The implant functions effectively throughout the follow-up period without major malfunctions, loosening, or breakage. Mechanical Failure is defined as reoperation with device removal related to the device implant loosening, implant fracture, repeated joint dislocation. Biological Failure is defined as reoperation with device removal related to the device periprosthetic infection, biofilm, allergic reaction to the implant materials.

SECONDARY OUTCOMES:
Safety endpoint: Occurrence rate of periprosthetic infection | From implantation up to 10-year follow-up, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal or re-intervention due to implant-related or non-implant-related complications.
  Periprosthetic infection is defined as a confirmed microbial infection involving the implanted TMJ prosthesis. After implantation, but in the long term, it could also contribute to a gradual decline in implant function over time, so a cure of the infection usually requires removal or replacement of the prosthesis.
  Unit of Measure: Percentage of participants (%): The occurrence rate will be calculated as the proportion of participants with at least one confirmed periprosthetic infection (numerator) divided by the total number of study participants (denominator).
Radiological Parameter Endpoint: Presence of Ectopic Bone | From implantation through 10-year follow-up, with (CB)CT scans performed at Week 1, Week 4, Year 1, Year 3, Year 5, and Year 10, or until device removal.
  The presence of ectopic bone refers to the formation of bony structures in locations where bone tissue is not typically found, including abnormal bone growth around the implant and changes in the shape or contour of surrounding bone structures. This is assessed by the investigator through radiological imaging. Additional information captured if present:
  Ectopic bone location: Soft tissue, Ramus, Joint space Shape/contour changes: Present, Absent Unit of Measure: Occurrence rate of ectopic bone.
Performance Endpoint: Mean Interincisal Opening (MIO) | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  The inter-incisal opening is the magnitude of the aperture formed between the upper and lower incisors during maximal mouth opening. It is commonly assessed by measuring the distance between the incisal edges of the upper and lower incisors. This metric is relevant in medical and dental evaluations as it estimates the mandibular range of motion and offers diagnostic insights into various orofacial conditions, including temporomandibular joint disorders and restricted jaw mobility.The reference values for MIO can vary among individuals and depend on factors such as age, gender, and overall health. Normal ranges typically fall between 35 to 55 mm. The amount of open bite should be subtracted for the MIO measurement, and in deep bites, the amount of vertical overlap should be added to the measurement for accurate determination of MIO. A larger MIO is considered as better.
The relationship between the device's success rate and the underlying medical condition | Up to 10-year follow-up post-implantation, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal due to mechanical or biological failure, stratified by underlying medical condition
  The relationship between the device's success rate and the underlying medical condition for up to 10 years could help in understanding how different medical conditions impact the success rate of the TMJ replacement device over time. It could highlight which conditions are associated with better or worse outcomes.
Mean implantation time | From implantation until device removal or up to 10-year follow-up post-implantation.
  Mean implantation time of the device from surgery until device removal or 10 years, if the device remains in place: Knowing the average duration the device remains in place before removal or up to 10 years can give an indication of the longevity of the device and how well it performs over time.
Surgical operation time | At procedure (intraoperative).
  Surgical operation time evaluates the efficiency of the surgical procedure and will be compared to virtual surgery planning vs. conventional surgeries. Also, it will be useful for potential areas for improvement in the surgical technique.
Total hospital post-operative stay | From surgery completion untill discharge date, when the patient is deemed clinically stable and released from hospital care, assessed up to 30 days post-operatively, with the duration varying based on underlying conditions and recovery progress.
  Total hospital post-operative stay (days) and its association with the underlying medical condition and the device: understanding the length of hospital stay post-surgery and its association with the underlying medical condition and the device can provide insights into recovery times, potential complications, and overall patient outcomes.
Perioperative complications | The perioperative period, encompassing the pre-operative (before surgery), intra-operative (during surgery), and post-operative (after surgery) phases, from patient admission for surgery until discharge home.
  Perioperative complications related and unrelated to the TMJ System, including allergic reaction to the anesthetic or titanium (anaphylaxis), complications related to the anesthesia, hematoma, or others.
Intraoperative blood loss (mL) | At procedure (intraoperative)
  Intraoperative blood loss is important for patient safety. Monitoring and analyzing this data can help optimize planning and surgical techniques to minimize blood loss and associated risks. Estimated blood loss by visual inspection or gravimetric method.
Technical success of the implantation | At procedure (intraoperative), and at first post-operative imaging (CB)CT at Week 1 for comparison with the pre-operative plan.
  Technical success of the implantation is defined by the surgeon and indicates whether the TMJ System was implanted according to the pre-operative plan.
  This is a binary question if technical success was achieved.
  For patients where technical success was not achieved, the following details will be captured:
  Nature of Device Problem: Design issues, surgical guide fit, TMJ trial implant, or other (specify).
  Surgical response: Adaptation, use of standard devices, or other (specify). Cause identification: Yes/No, with details if Yes.
  Consequences: None, life-threatening injury, permanent impairment, prolonged hospitalization, increased intervention time, new surgery, or other (serious or not).
  Device Deficiency: Could have led to a serious adverse device effect (SADE)? Yes/No/Unknown.
  Unit of Measure: rate of technical success, expressed as the percentage of successful implantations across all patients, with breakdowns for issues that led to a lack of success.
Radiological Parameter Endpoint: Displacement of Ramus Component | From implantation through 10-year follow-up, with (CB)CT scans performed at Week 1, Week 4, Year 1, Year 3, Year 5, and Year 10, or until device removal.
  Displacement of the ramus component, evaluated by the investigator, will be assessed using (cone beam) computed tomography scans. The outcome is binary: displacement is either "Yes" or "No." In cases of displacement, additional information such as condylar position relative to the fossa, articular eminence, glenoid fossa, articular disc, or condylar translation or rotation will be captured.
  Unit of Measure: Percentage of participants with ramus component displacement.
Safety endpoint: Occurrence rate of weakness of the temporal branch of the facial nerve | From implantation up to 10-year follow-up, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal or re-intervention due to implant-related or non-implant-related complications.
  Postoperative weakness of the temporal branch of the facial nerve is defined as a reduction or loss of motor function affecting the frontalis or orbicularis oculi muscles, observed clinically through facial asymmetry, reduced forehead movement, or brow ptosis. Assessment will be performed according to the site's standard of care practice, for example via standardized facial nerve function grading (e.g., House-Brackmann scale or clinical neurological exam).
  Unit of Measure: Percentage of participants (%). The occurrence rate will be calculated as the proportion of participants with clinically confirmed weakness of the temporal branch of the facial nerve (numerator) divided by the total number of study participants (denominator).
Safety endpoint: Occurrence rate of marginal mandibular palsy | From implantation up to 10-year follow-up, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal or re-intervention due to implant-related or non-implant-related complications.
  Marginal mandibular palsy is defined as partial or complete loss of motor function of the lower lip muscles. Assessment will be performed through clinical examination according to the site's standard of care, e.g. graded using the House-Brackmann scale or similar facial nerve evaluation protocol.
  Unit of Measure: Percentage of participants (%). The occurrence rate will be calculated as the proportion of participants with clinically confirmed marginal mandibular branch palsy (numerator) divided by the total number of study participants (denominator).
Safety endpoint: Occurrence rate of total facial palsy | From implantation up to 10-year follow-up, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal or re-intervention due to implant-related or non-implant-related complications.
  Total facial palsy refers to complete or near-complete loss of motor function across all branches of the facial nerve on the affected side, typically resulting in inability to raise the eyebrow, close the eye, or move the mouth on that side. Diagnosis will be based on clinical neurological examination according to the site's standard of care, e.g. graded using the House-Brackmann scale or equivalent validated facial nerve grading system.
  Unit of Measure: Percentage of participants (%). The occurrence rate will be calculated as the proportion of participants with clinically confirmed total facial nerve palsy (numerator) divided by the total number of study participants (denominator).
Safety endpoint: Occurrence rate of other sensory changes (lip, tongue, auriculotemporal nerve) | From implantation up to 10-year follow-up, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal or re-intervention due to implant-related or non-implant-related complications.
  Sensory changes refer to altered or diminished sensation in areas innervated by branches of the trigeminal nerve, including the lower lip, tongue, and auriculotemporal region. These may present as numbness, tingling, hypoesthesia, or dysesthesia, and will be assessed through patient-reported symptoms and clinical neurological examination (e.g., light touch and pinprick testing), according to the site's standard of care.
  Unit of Measure: Percentage of participants (%). The occurrence rate will be calculated as the proportion of participants with one or more confirmed sensory changes involving the lip, tongue, or auriculotemporal nerve (numerator) divided by the total number of study participants (denominator).
Safety endpoint: Occurrence rate of other general post-operative complications | Starting after operation, up to 10-year follow-up, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal or re-intervention due to implant-related or non-implant-related complications.
  Other general post-operative complications include any adverse events not otherwise categorized,. These events will be recorded and classified according to their nature, severity, and relation to the implant procedure, as assessed by the investigator according to the site's standard of care.
  Unit of Measure: Percentage of participants (%). The occurrence rate will be calculated as the proportion of participants experiencing at least one general post-operative complication (numerator) divided by the total number of study participants (denominator).
Safety endpoint: Occurrence rate of stable implant components | From implantation up to 10-year follow-up, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal or re-intervention due to implant-related or non-implant-related complications.
  Stable implant components refer to the retention and proper function of the TMJ implant components, including the plate, screws, and prosthesis, without evidence of loosening, fracture, or migration. The assessment will include clinical examination and radiographic imaging (e.g., X-rays, CT scans), conducted according to the site's standard of care.
  Unit of Measure: Percentage of participants (%). The occurrence rate will be calculated as the proportion of participants with stable implant components (no loosening, fracture, or migration) (numerator) divided by the total number of study participants (denominator).
Safety endpoint: Re-intervention rate up to 10 years follow-up, implant-related or not. | After implantation up to 10-year follow-up, with evaluations at Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal or re-intervention due to implant-related or non-implant-related complications.
  Re-intervention due to implant-related or non-implant-related complications. Unit of Measure: Percentage of participants (%) The re-intervention rate will be calculated as the proportion of participants who undergo re-intervention (numerator) divided by the total number of study participants (denominator).
Performance Endpoint: Occlusion | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  Angle's classification of malocclusion is a widely recognized system used to categorize dental occlusions based on the relationship between the first molars and the canines. This classification divides malocclusions into three primary categories: Class I, where the first molar relationship is normal but other dental discrepancies may exist; Class II, characterized by a retrognathic relationship of the first molars, often accompanied by overbite; and Class III, where the first molars are positioned more mesially, leading to an underbite. The classification is performed through clinical examination, where the occlusal relationships are assessed, typically using dental casts or intraoral assessments to evaluate the alignment and positioning of the teeth.
Performance Endpoint: Dentition | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  Dental status will be recorded as: Edentulous, Complete dentition, or Partial dentition. In the case of partial dentition, missing teeth will be recorded individually using the Fédération Dentaire Internationale (FDI) tooth numbering formula.
Performance Endpoint: Diet Consistency Evaluation Numerical Rating Scale (NRS) | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  Before and after surgery, the evaluation of diet consistency is essential to assess the patient's ability to chew and swallow different types of food, as well as to measure subjective diet limitations. Each participant will undergo a diet consistency evaluation prior to and following surgery. The participants will be asked to indicate which of the following options applies to their diet:
  0 = no restrictions at all - normal diet 10 = liquids only
Performance Endpoint: Speech Numerical Rating Scale (NRS) | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  Speech scores will be measured by a Numerical Rating Scale (NRS) ranging from 0 to 5, where 0 represents no function and 5 represents optimal condition. This evaluation will assess the patient's ability to speak comfortably and clearly following the temporomandibular joint implant surgery. The assessment will be conducted at baseline, discharge, and during all follow-up visits to track any improvements or limitations in speech.
Performance Endpoint: Jaw Function Numerical Rating Scale (NRS) | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  The Jaw Function Numerical Rating Scale (NRS) is an 11-point scale used to measure subjective jaw function. The endpoints of the scale represent the extremes of jaw mobility, where 0 indicates normal jaw movement and 10 indicates no jaw movement. This evaluation captures the patient's perception of their functional jaw ability following temporomandibular joint implant surgery and throughout the follow-up period.
Performance Endpoint: Oral Health Impact Profile-14 (OHIP-14) | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  The Oral Health Impact Profile-14 (OHIP-14) is a validated 14-item questionnaire used to assess oral health-related quality of life by measuring the frequency of problems across seven domains, including functional limitation, physical pain, psychological discomfort, and social disability. Responses are rated on a Likert-type scale from 0 (never) to 4 (very often), with higher scores indicating greater impact on daily life.
Performance Endpoint: EuroQoL 5-Dimension 5-Level (EQ-5D-5L) | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  The EuroQoL 5-Dimension 5-Level (EQ-5D-5L) is a standardized questionnaire used to assess health-related quality of life across five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-each with five severity levels. It also includes a visual analog scale (EQ VAS) where patients rate their overall health from "the worst" to "the best health you can imagine." Higher values on the EQ VAS and lower dimension scores indicate better perceived health status.
Performance Endpoint: Helkimo Clinical Dysfunction Index | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  The Helkimo Clinical Dysfunction Index is a simple and quick test that aids in evaluating key factors such as pain, joint sounds, mandibular mobility, and muscle function to provide a comprehensive understanding of the severity of TMJ dysfunction. It is important to note that while the Helkimo Clinical Dysfunction Index can help assess and evaluate TMJ dysfunction, it is not directly associated with TMJ replacement procedures. From question A to E, 3 options can be chosen with a corresponding value of 0, 1 or 5, where a higher value relates to worse clinical symptoms. These are then summated to categorise the patient in a dysfunction group (range from symptom free to severe dysfunction).
Performance Endpoint: Patient Satisfaction Numeric Rating Scale (NRS) - Functional and Aesthetic | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  The Patient Satisfaction Numeric Rating Scale (NRS) is a single-item, 11-point scale used to assess the patient's satisfaction with functional and aesthetic outcomes of the surgical procedure. Scores range from 0 (no satisfaction) to 10 (complete satisfaction), with higher scores indicating greater satisfaction.
Performance Endpoint: Surgeon Satisfaction Numeric Rating Scale (NRS) - Functional and Morphological/Aesthetic | From baseline (pre-implantation) through 10-year follow-up post-implantation, with evaluations at baseline, discharge, Week 1, Week 4, Month 3, Month 6, Year 1, Year 2, Year 3, Year 5, and Year 10, or until device removal.
  The Surgeon Satisfaction Numeric Rating Scale (NRS) is a single-item, 11-point scale used to assess the surgeon's satisfaction with the functional and morphological/aesthetic outcomes of the surgical procedure. Scores range from 0 (not satisfied) to 10 (completely satisfied), reflecting the surgeon's evaluation of key aspects such as preoperative planning, intraoperative performance, and postoperative outcomes.
Radiological Parameter Endpoint: Fracture of Ramus Component | From implantation through 10-year follow-up, with (CB)CT scans performed at Week 1, Week 4, Year 1, Year 3, Year 5, and Year 10, or until device removal.
  Fracture of the ramus component, evaluated by the investigator, will be assessed using (cone beam) computed tomography scans. The outcome is binary: fracture is either "Yes" or "No." If a fracture is detected, additional descriptive details will captured such as bone discontinuity or interruption, presence of bone fragments or displacement of bone fragments, and changes in alignment or angulation.
  Unit of Measure: Percentage of participants with ramus component fracture.
Radiological Parameter Endpoint: Screw Loosening | From implantation through 10-year follow-up, with (CB)CT scans performed at Week 1, Week 4, Year 1, Year 3, Year 5, and Year 10, or until device removal.
  Screw loosening will be evaluated by the investigator using (cone beam) computed tomography scans and reported as a binary outcome (present or not present). For cases where loosening is observed, additional details such as a visible gap between the screw and bone surface, change in screw position, or the presence of radiolucent lines around the screws (indicating potential movement) will be captured.
  Unit of Measure: Occurrence rate (%)
Radiological Parameter Endpoint: Bone Resorption or Osteolysis Around the Implant | From implantation through 10-year follow-up, with (CB)CT scans performed at Week 1, Week 4, Year 1, Year 3, Year 5, and Year 10, or until device removal.
  Bone resorption or osteolysis of the surrounding bone will be evaluated by the investigator using (cone beam) computed tomography scans. The presence or absence of resorption or osteolysis will be recorded as a binary outcome. If present, additional information will be captured, including thinning of bone around the implant, presence of radiolucent areas indicating bone loss, changes in the shape or contour of bone structures, and any progressive decrease in bone density around the implant components.
  Unit of Measure: Occurrence rate (%)
Radiological Parameter Endpoint: Status of Bone Grafts (if used) | From implantation through 10-year follow-up, with (CB)CT scans performed at Week 1, Week 4, Year 1, Year 3, Year 5, and Year 10, or until device removal.
  The status of bone grafts (if used) will be evaluated by the investigator through (cone beam) computed tomography scans. The assessment will capture the following:
  Integration with native bone: Well Integrated, Partially Integrated, Not Integrated Density of graft material: Normal, Decreased, Increased Volume of graft material: Stable, Decreased, Increased Unit of measurement: rate of occurrence for each of the graft material statuses (e.g., well integrated, partially integrated, not integrated, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No